CLINICAL TRIAL: NCT04885309
Title: Efficacy and Safety of Obturator Nerve Block During Transurethral Resection on Non-muscle Invasive Intermediate and High Risk Lateral Wall Bladder Tumours Comparing Nerve Stimulator-guided Obturator Nerve Block With Spinal Anaesthesia and Spinal Anaesthesia: A Prospective Randomized Controlled Study
Brief Title: Efficacy and Safety of Obturator Nerve Block During Transurethral Resection on Non-muscle Invasive Intermediate and High Risk Lateral Wall Bladder Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yıldız, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONB2021
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Bladder Cancer Stage 0; Bladder Cancer Stage I
Keywords: Non-muscle invasive bladder cancer; Obturator nerve block; Transurethral resection
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obturator Nerve Block + Spinal Anaesthesia (Active Comparator): Patients who underwent obturator nerve block with spinal anesthesia prior to TURBT
  Interventions: Procedure: Nerve Stimulator-guided Obturator Nerve Block
- Spinal Anaesthesia (Sham Comparator): Patients who underwent spinal anesthesia prior to TURBT
  Interventions: Procedure: Nerve Stimulator-guided Obturator Nerve Block

INTERVENTIONS:
Procedure: Nerve Stimulator-guided Obturator Nerve Block — Following the confirmation of spinal anesthesia level in the patients in the ONB group while in the lithotomy position, ONB was applied unilaterally or bilaterally, depending on the tumor position. A needle with a nerve stimulator was advanced vertically 2 cm below and 2 cm from the pubic tubercle. The needle is inserted through the skin and into the lower ramus of the pubic bone. When contraction was observed in the adductor muscle groups and the aspiration was negative, 10 mL 0.25% levobupivacaine at 0.3-0.5 mA was administered. The operation was started 10 minutes after the injection. TURBT operations were performed with a 30 degree optic and a 26 F bipolar resectoscope. All spinal anesthesia and ONB procedures were performed by the same anesthesia team. All TURBT operations were performed by the same surgeon.

SUMMARY:
In this prospective randomized controlled study, the effects of obturator nerve block (ONB) on obturator reflex, incomplete resection, perforation, tumor recurrence and progression, presence of muscle tissue in the specimen, need for second transurethral resection of bladder tumours (TURBT) and postoperative complications were investigated in patients who underwent TURBT for intermediate and high risk lateral wall non-muscle invasive bladder tumours (NMIBC).

DETAILED DESCRIPTION:
Bladder cancer is among the ten most common types of cancer in the world, with about 550,000 new cases per year. According to GLOBOCAN (Global Cancer Incidence, Mortality and Prevalence) data, bladder cancer accounts for 3% of cancer diagnoses worldwide. It is more common, especially in developed countries. A total of 90% of bladder cancer diagnoses are made in people 55 years of age or older, and the disease is four times more common in men than in women. NMIBC are divided into four groups as low-medium-high and very high risk according to EORTC (European Organization for Research and Treatment of Cancer). Early recurrence was reported as 15%, late recurrence as 25% and progression as 9% with BCG treatment in medium and high risk NMIBC. TURBT is the basic approach in diagnosis and treatment.

The obturator nerve passes through the obturator foramen of the pubis and innervates the adductor muscles of the thigh. It lies within the pelvic cavity close to the prostatic urethra, bladder neck and inferolateral bladder wall. In TURBT, when the bladder is filled with irrigation fluid, the obturator nerve is very close to the bladder sidewall. While performing TURBT of lateral wall bladder tumors, neighboring obturator nerve stimulation may occur during surgical resection, resulting in adductor contraction and leg jerking. This condition, called the obturator reflex, occurs between 55.3% and 100% of lateral bladder tumors.

Serious complications can occur in TURBT, one of which is bladder perforation that may require laparotomy and open repair. Perforation is also associated with poor patient outcomes due to the spread of the tumor into the abdominal cavity and the inability to apply single immediate instillation of intravesical chemotherapy. One of the most important factors affecting the success of TURBT is the presence of residual tumor as a result of incomplete resection. Incomplete resection is associated with both general recurrence and particularly local recurrence, as well as shortening disease-free survival. One of the most important indicators of complete resection is the presence of the detrusor muscle in the TURBT specimen. However, in 10% of all cases, it has been reported that there is no detrusor muscle tissue in the TURBT specimen. Various methods such as administration of muscle relaxants under general anesthesia, less filling of the bladder, reduction of electric current, using a 90-degree classical loop, using bipolar plasmakinetic energy and performing tumor resection with small pieces have been proposed in order to prevent the failure and complications due to obturator reflex that may occur in TURBT.

In combination with spinal anesthesia, ONB is one of the most effective methods used to inhibit the obturator reflex. The importance of spinal anesthesia has increased especially due to the COVID-19 outbreak. Surgery under local / regional anesthesia is recommended as much as possible, especially during the pandemic process, compared to general anesthesia. In this way, it is aimed to reduce the risk of aerosol generating procedures and subsequent viral transmission. ONB has gained more importance in recent years as a result of being performed together with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Lateral wall intermediate and high risk non-muscle invasive bladder cancer

Exclusion Criteria:

* Low risk non-muscle invasive bladder cancer
* Contraindications for spinal anesthesia
* History of allergy to local anesthetic agents
* Coagulopathy
* Neuromuscular diseases affecting the central nervous system
* Obturator nerve injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of Obturator Reflex | One year
  Rate of patients who had an obturator reflex during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No